CLINICAL TRIAL: NCT03572790
Title: The Effect of Seven Day Prucalopride Administration on Emotional Processing in Healthy Volunteers
Brief Title: Effects of Seven Day Prucalopride Administration in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, drsusannahmurphy, Senior Research Fellow, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pruc_7d
Record Dates: First submitted 2018-06-07; First posted 2018-06-28 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Molecular Mechanisms of Pharmacological Action; Depression; Depressive Disorder; Mood Disorders; Mental Disorders; Antidepressive Agents; Cognition
Keywords: 5-HT4; Prucalopride; Resolor; Functional Magnetic Resonance Imaging (fMRI); Emotional Processing; Healthy Volunteers
MeSH Terms: conditions — Depression; Depressive Disorder; Mood Disorders; Mental Disorders | interventions — prucalopride

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of two groups (prucalopride or placebo). Participants in the prucalopride group will receive 1mg once daily for seven days. Participants in the placebo group will receive a lactose placebo once daily for seven days. Note that the study is not assessing the safety or efficacy of prucalopride, rather it is using prucalopride to assess the behavioural and neural effects of 5-HT4 partial agonists.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prucalopride (Experimental)
  Interventions: Drug: Prucalopride
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Prucalopride — 1mg prucalopride capsule, once daily for seven days
  Other Names: Resolor
  Arms: Prucalopride
Other: Placebo — Lactose placebo capsule, once daily for seven days
  Arms: Placebo

SUMMARY:
This study will investigate whether seven days administration of the serotonin receptor subtype 4 (5-HT4) partial agonist prucalopride has effects on emotional processing and neural activity in healthy volunteers, compared to placebo administration. Using an experimental medicine approach, the effects of prucalopride on cognitive biomarkers of antidepressant action will be characterised. In a double-blind design, participants will be randomised to receive seven days administration of either prucalopride (1mg daily) or placebo. All participants will come for a Screening visit, Research Visit One (including an MRI scan) and Research Visit Two (including measures of emotional processing and non-emotional cognition). The primary study hypothesis is that seven-day prucalopride administration will have positive effects on emotional processing and reward sensitivity. A secondary hypothesis is that seven-day prucalopride administration will alter non-emotional cognition. Finally, the study will test the hypothesis that seven day prucalopride administration will alter neural activity during an emotional faces task and a memory task.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or female
* Aged 18-40 years
* Sufficiently fluent English to understand and complete the task
* Right handed
* Body Mass Index in the range of 18-30
* Not currently taking any medications (except the contraceptive pill)

Exclusion Criteria:

* Not fluent in English
* Any past or current Axis 1 DSM-V psychiatric disorder
* Current usage of psychoactive medication (except the contraceptive pill, the Depo-Provera injection or the progesterone implant)
* Current usage of any medication that will influence the MRI scan
* Current or past history of drug or alcohol dependency
* Currently pregnant or breastfeeding
* Study visits due to take place during the pre-menstrual week (female participants asked details of their menstrual cycle to schedule the study outside this week)
* Not right handed
* Body Mass Index outside the range of 18-30
* History of cardiac, thyroid, or liver problems
* An autoimmune disorder
* Current, or a history of, gastro-intestinal disorder or irritable bowel syndrome
* Epilepsy
* Known lactate deficiency or any other problem absorbing lactose, galactose, or glucose
* Participation in a study which uses the same computer tasks as those used in the present study
* Participation in a study that involves the use of a medication within the last three months
* Smoker > 5 cigarettes per day
* Typically drinks > 6 caffeinated drinks per day
* Any contraindication to MRI scanning (e.g. metal objects in the body, pacemakers, significant claustrophobia)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Recognition of positive and negative facial expressions | Completed on Day 7
  Accuracy to recognise positive and negative facial expressions (anger, disgust, fear, happy , sad, surprise)
Performance on Auditory Verbal Learning Task (AVLT) | Completed on Day 7
  Accuracy on AVLT (number of items recalled across blocks)

SECONDARY OUTCOMES:
Neural response to emotional faces | Completed on Day 6
  Blood Oxygen Level Dependent (BOLD) signal in a network including the amygdala, anterior cingulate cortex, and orbitofrontal cortex
Neural response to novel vs repeated scenes | Completed on Day 6
  BOLD signal to scenes that have previously been seen compared to novel scenes in a network including the hippocampus and parahippocampal regions
Reward sensitivity | Completed on Day 7
  Sensitivity to reward as measured by the Probabilistic Instrumental Learning Task (PILT)
Categorisation, recall, and recognition of emotional words | Completed on Day 7
  Accuracy and reaction time to categorise positive and negative descriptor words; number of words correctly (hits) and incorrectly (false alarms) recalled and recognised
Vigilance to fearful and happy faces on the Facial Dot Probe Task (FDOT) | Completed on Day 7
  Vigilance derived from reaction time
Resting state connectivity | Completed on Day 6
  Resting state connectivity (using resting state fMRI) including the default mode network, salience network, affective network, and limbic system, identified via correlations between spontaneous BOLD activity in spatially independent regions while participants are not actively engaged in an experimental task
Relative and global cerebral blood flow | Completed on Day 6
  Arterial spin labelling (ASL) global and cerebral blood flow
Visual short term memory on the Oxford Memory Test (OMT) | Completed on Day 7
  Proportion of correct probe selections, absolute error for probe location, reaction time, and proportion of misbinding errors

CONTACTS AND LOCATIONS:
Overall Officials: Susannah E Murphy, DPhil, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Cates AN, Martens MAG, Wright LC, Gibson D, Spitz G, Gould van Praag CD, Suri S, Cowen PJ, Murphy SE, Harmer CJ. 5-HT4 Receptor Agonist Effects on Functional Connectivity in the Human Brain: Implications for Procognitive Action. Biol Psychiatry Cogn Neurosci Neuroimaging. 2023 Nov;8(11):1124-1134. doi: 10.1016/j.bpsc.2023.03.014. Epub 2023 Apr 23. PMID 37098409
- See also: Psychopharmacology and Emotion Research Laboratory — http://www.perloxford.org

DOCUMENTS (3):
  • Study Protocol (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT03572790/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT03572790/SAP_004.pdf
  • Informed Consent Form (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT03572790/ICF_001.pdf